CLINICAL TRIAL: NCT00513019
Title: A Double-Blind Study of Lamictal in Neurotic Excoriation
Brief Title: Double-Blind Lamictal (Lamotrigine) in Neurotic Excoriation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0703M03384
Record Dates: First submitted 2007-08-07; First posted 2007-08-08 (Estimated); Results first posted 2013-09-27 (Estimated); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Neurotic Excoriation; Pathologic Skin Picking; Psychogenic Excoriation; Dermatillomania
Keywords: Neurotic Excoriation; Pathologic Skin Picking; Psychogenic Excoriation
MeSH Terms: conditions — Excoriation Disorder | interventions — Lamotrigine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Lamictal (lamotrigine)
  Interventions: Drug: Lamictal (lamotrigine)
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lamictal (lamotrigine) — once daily from beginning to end of study. Dosage varies.
  Other Names: lamotrigine
  Arms: 1
Drug: Placebo — daily
  Arms: 2

SUMMARY:
The goal of the proposed study is to evaluate the comparative efficacy of Lamictal (lamotrigine) to placebo in neurotic excoriation. Thirty subjects with neurotic excoriation will receive 12 weeks of double-blind treatment with Lamictal (lamotrigine) or matching placebo. The hypothesis to be tested is that Lamictal (lamotrigine) will be more effective than placebo in patients with neurotic excoriation. The proposed study will provide needed data on the treatment of a disabling disorder that currently lacks a clearly effective treatment.

DETAILED DESCRIPTION:
The study will consist of 12 weeks of double-blind treatment with Lamictal (lamotrigine) compared to placebo (1:1) in 30 subjects with neurotic excoriation.

ELIGIBILITY:
Inclusion Criteria:

1. men and women age 18-65;
2. current diagnosis of neurotic excoriation.

Exclusion Criteria:

1. unstable medical illness or clinically significant abnormalities on prestudy laboratory tests or physical examination;
2. history of seizures;
3. myocardial infarction within 6 months;
4. current pregnancy or lactation, or inadequate contraception in women of childbearing potential;
5. a need for medication other than Lamictal with possible psychotropic effects or unfavorable interactions with Lamictal;
6. clinically significant suicidality;
7. lifetime history of DSM-IV bipolar disorder type I, dementia, or schizophrenia or any other DSM-IV psychotic disorder;
8. current or recent (past 3 months) DSM-IV substance abuse or dependence;
9. illegal substance use within 2 weeks of study initiation;
10. initiation of psychotherapy or behavior therapy from a mental health professional within 3 months prior to study baseline;
11. previous treatment with Lamictal (lamotrigine);
12. treatment with investigational medication or depot neuroleptics within 3 months, with fluoxetine within 6 weeks, or with other psychotropics within 2 weeks prior to study baseline;
13. current treatment with an anti-epileptic medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-08; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon E Grant, M.D., Principal Investigator — University of Minnesota
Locations (1):
- Ambulatory Research Center, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: August 2007 - July 2009
Groups:
- Lamictal: The subjects began lamotrigine at 25 mg/d every other day for 1 week. At week 1, the dose was raised to 25 mg/d. At week 2, the dose was raised to 50 mg/d for 2 weeks. Thereafter, all visits were scheduled every 2 weeks at which times the dose could be increased to 100 mg/d, then 200 mg/d, and finally 300 mg/d unless clinical improvement was attained at a lower dose (clinical improvement was assessed by the investigator with respect to skin picking behavior, thoughts, and urges).
- Placebo: Placebo pills (identical to lamictal pills) were taken by mouth once daily.
Period: Overall Study
Arm/Group | Lamictal | Placebo
Started | 17 | 18
Completed | 12 | 13
Not Completed | 5 | 5
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lamictal | Placebo | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 18 | 35
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (14.1) | 31.6 (13.3) | 32.8 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 17 | 18 | 35

OUTCOME MEASURES:

1. Primary Outcome: The Yale-Brown Obsessive Compulsive Scale Modified for Neurotic Excoriation (NE-YBOCS) Will be the Primary Outcome Measure
Description: The Yale-Brown Obsessive Compulsive Scale Modified for Neurotic Excoriation (NE-YBOCS) was the primary outcome measure - severity of illness. The NE-YBOCS is a reliable and valid, 10-item, clinician-administered scale that rates buying symptoms within the last seven days, on a severity scale from 0 to 4 for each item (total scores range from 0 to 40 with higher scores reflecting greater illness severity).
Time Frame: beginning and at each visit until the end of their participation in the study (12-weeks); investigator rated. Note: Reported mean and standard deviation is the final reported data point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lamictal | Placebo
Number analyzed (Participants) | 17 | 18
units on a scale | 15.25 (4.1) | 16.13 (3.6)

ADVERSE EVENTS:
Arm/Group | Lamictal | Placebo
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 1/17 | 0/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Lamictal (N=17) | Placebo (N=18)
Disorientation (Psychiatric disorders) | 1/16 (1) | 0/16 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No